CLINICAL TRIAL: NCT07130903
Title: A Phase 2 Study of Amplitude-Modulated Radiofrequency Electromagnetic Fields (AM RF EMF) in Combination With Fruquintinib in Refractory Metastatic Colorectal Cancer
Brief Title: Amplitude-Modulated Radiofrequency Electromagnetic Fields (AM RF EMF) in Combination With Fruquintinib in Refractory Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: THERABIONIC INC. (Other)
Responsible Party: Principal Investigator, Mohammed Najeeb Al Hallak, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-035
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Adenocarcinoma
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Amplitude-modulated radiofrequency electromagnetic fields device plus Fruquintinib (Experimental): TheraBionic P1 amplitude-modulated radiofrequency electromagnetic fields device 3 times daily (continuous) plus Fruquintinib daily (3 weeks on and 1 week off)
  Interventions: Drug: Fruquintinib; Device: TheraBionic P1

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib is a small molecule tyrosine kinase inhibitor (TKI) that targets VEGFR-1, -2, and -3, with a novel chemical structure which belongs to the quinazoline class
  Other Names: Fruzaqla; HMPL-013
Device: TheraBionic P1 — TheraBionic P1 is a amplitude-modulated radiofrequency electromagnetic fields (AM RF EMF) device

SUMMARY:
The goal of this clinical trial is to learn if adding amplitude-modulated radiofrequency electromagnetic fields (AM RF EMF) to Fruquintinib in metastatic colorectal cancer that has not responded to other standard treatment is:

* Effective in improving survival
* safe and tolerable

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed metastatic colorectal adenocarcinoma. There must be previous documentation of RAS (Rat sarcoma mutation), BRAF (B-Raf proto-oncogene, Serine/threonine kinase), MSI/MMR (microsatellite instability, mismatch repair) , and HER2 (Human epidermal growth factor receptor 2) status.
* Participant must have progressed on or been intolerant to the following previous treatments (if not contraindicated):

  * Fluoropyrimidine-, oxaliplatin-, or irinotecan-based chemotherapy
  * Anti-VEGF (vascular endothelial growth factor) biological therapy, such as bevacizumab, aflibercept, or ramucirumab
  * If RAS is wild type, an anti-EGFR (epidermal growth factor receptor) therapy like cetuximab or panitumumab
* Participant must have evaluable disease as defined by the investigator using CT (computed tomography), MRI (magnetic resonance imaging), or PET (positron emission tomograph) scan.
* Participant must have a body weight ≥ 40 kg.
* Participant must be aged 22 years or older.
* Participant must be able to understand a written informed consent document and be willing to sign it.
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Participant must have adequate organ and marrow function within 14 days prior to the initiation of treatment as described below:
* Participant should have an expected lifespan of >12 weeks as determined by the investigator.
* Fruquintinib is suspected to cause loss of human pregnancy and impaired development of the embryo or fetus. Therefore, women of child-bearing potential must agree to avoid becoming pregnant and male participants should avoid impregnating a female partner starting at initiation of treatment up until at least 14 days after the last fruquintinib dose.

Exclusion Criteria:

* Participants with uncontrolled hypertension per investigator discretion.
* Participants with a history or presence of gastric/duodenal ulcer or ulcerative colitis, hemorrhage of an unresected gastrointestinal tumor, perforation, fistulas, or any other condition that could, in the investigator's judgment, result in gastrointestinal hemorrhage or perforation.
* Participants with a history or presence of hemorrhage from any other site (i.e., lower GI bleed, hemoptysis or hematemesis) within two months prior to screening.
* Participants with a history of a thromboembolic event, including deep vein thrombosis (DVT), pulmonary embolism (PE), or arterial embolism within three months prior to screening unless they are on a stable dose of anticoagulant and no further evidence of active thromboses are seen on CT scan or venous Doppler imaging. Participants with saddle (massive) pulmonary embolism that require thrombectomy/thrombolysis within 12 months of screening are excluded from the trial.
* Participants with a history of stroke and/or transient ischemic attack within 12 months prior to screening.
* Participants with clinically significant cardiovascular disease, including but not limited to acute myocardial infarction or coronary artery bypass surgery within six months prior to enrollment, severe or unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, ventricular arrhythmias requiring treatment, or previous left ventricular ejection fraction (LVEF) < 50% by echocardiogram.
* Participants with corrected QT interval using the Fridericia method (QTcF) > 480 msec or any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in a first-degree relative.
* Participants taking concomitant medications with a known risk of causing QT prolongation and/or torsades de pointes. (Source list is continuously updated online at www.crediblemeds.org.)
* Participants taking systemic anti-neoplastic therapies four weeks prior to the first dose of study drug, including chemotherapy, biotherapy, or immunotherapy. Palliative radiation is allowed if it does not cover all evaluable disease.
* Participants taking systemic small molecule targeted therapies (e.g., tyrosine kinase inhibitors) within five half-lives or four weeks, whichever is shorter, prior to the first dose of study drug.
* Participants who have undergone major surgery within 30 days prior to the first dose of study drug or if they still have unhealed surgical incision from previous surgery.
* Participants with any unresolved toxicities from a previous antitumor treatment greater than NCI CTCAE v5.0 grade 2.
* Participants that have current drug or alcohol abuse.
* Participants with known human immunodeficiency virus (HIV) infection are not eligible if their viral load and/or CD4 (cluster of differentiation 4) count are considered poorly controlled with anti-HIV therapy.
* Participants with a known history of active viral hepatitis. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Participants that test positive for hepatitis C virus (HCV) but are currently being treated are eligible if they have an undetectable HCV viral load.
* Participants with clinically uncontrolled active infections requiring intravenous antibiotics.
* Participants with tumor invasion of a large vascular structure (e.g., pulmonary artery, superior or inferior vena cava).
* Participants with brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy and without clinical imaging evidence of stable disease for 14 days or longer.
* Participants with known active secondary malignancy, unless, in the opinion of the investigator, it is unlikely to interfere with the safety and efficacy of the endpoints.
* Participants that are unable to take medication orally including those with dysphagia or an active gastric ulcer resulting from previous surgery (e.g., gastric bypass) or severe gastrointestinal disease, or any other condition that the investigator believes may affect absorption of fruquintinib.
* Participants with metabolic disorder that the investigator suspects may prohibit fruquintinib action, affect interpretation of study results, or put the participant at undue risk of harm based on the investigator's assessment.
* Participants that have received prior fruquintinib treatment.
* Participants with a known hypersensitivity to fruquintinib or any of its inactive ingredients including the azo dyes tartrazine, FD&C yellow 5, and sunset yellow FCF.
* Participants taking strong inducers or inhibitors of CYP3A4 within five half-lives or four weeks, whichever is longer, before the first dose of study drug. Refer to Appendix 2 for a comprehensive list of excluded medications related to CYP3A4.
* Participants that are taking any other investigational drugs.
* Participants with active oral mucosal inflammation, ulceration, or other pathology that could interfere with the use of TheraBionic P1 device (for example: mucositis, thrush, bleeding mucosal lesions, oral herpes, aphthous stomatitis, mouth ulcers, chancre sores, gingivostomatitis, herpangina, aphthae).
* Participants receiving calcium channel blockers and any agent blocking L-type or T-type voltage gated calcium channels (for example: amlodipine, nifedipine, ethosuximide, ascorbic acid/vitamin C, etc.) unless these drugs are discontinued at least 7 days prior to starting TheraBionic P1 device treatment. Participant must agree to abstain from using calcium channel blockers for the duration of treatment on study. Refer to Appendix 3 for a comprehensive list of excluded medications related to calcium channels.
* Participants that are pregnant or breastfeeding are ineligible for this study. If a breastfeeding participant would like to be part of this study, breastfeeding must be discontinued.
* Participants who have received a live vaccine ≤ 28 days before the first dose of fruquintinib. (Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.)
* Participants that do not agree to be followed according to the study protocol or have cognitive or physical inability to use the device.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-04-17 (Estimated); Study Completion 2030-04-17 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From start of treatment to 5 years after treatment discontinuation or death, whichever comes first
  Overall survival (OS) is defined as the time duration from treatment start until death of any cause. The distribution of OS will be graphically summarized by a Kaplan-Meier (KM) curve, and median OS (mOS) and its one-sided 85% (i.e., two-sided 70%) confidence interval (CI) will be estimated using KM estimates.

SECONDARY OUTCOMES:
Safety and Tolerability | From start of treatment to 28 days post device discontinuation
  Analyses will be performed for all participants who have received fruquintinib and TheraBionic P1 treatment. AEs will be graded based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. Adverse Events will be summarized by count and frequency. Corresponding two-sided 95% CI will be calculated using Clopper and Pearson's method.
Progression-free survival (PFS) | From start of treatment to 5 years after treatment discontinuation or death, whichever comes first
  Progression-free survival (PFS) is defined as the time duration from treatment start to progression or death of any cause. Progression of disease will be assessed and determined by the treating investigator. A one-sample log-rank test will be performed to evaluate PFS. The distribution of PFS will be graphically summarized by Kaplan-Meier (KM) curve and median PFS (mPFS) and its 95% CI will be estimated using KM estimates.
Rates of progressive disease | From start of treatment to 5 years after treatment initiation or death, whichever comes first
  The proportions of participants whose disease has progressed after treatment initiation will be computed by dividing the number of participants with progression by the total number of patients who were followed.
Changes in serum Carcinoembryonic Antigen (CEA) | Through study completion, up to 1 year
  Serum CEA will be measured at baseline, on Day 1 of each cycle, and at the end of treatment. Distribution of levels of serum CEA will be checked and, if needed, data transformation will be employed for normality. The levels of serum CEA will be descriptively summarized using mean, median, standard deviation (SD), range, and 95% CI per each time point. The changes in serum CEA will be also descriptively summarized using the same descriptive statistics. The associations between the change of serum CEA and each of efficacy outcomes will be descriptively evaluated using logistic and Cox proportional hazard regression models. The proportional hazard assumption will be checked and, if violated, a weighed Cox regression model or restricted mean survival time will be utilized.
Changes in serum microRNA (miRNA) | Through study completion, up to 1 year
  Serum miRNA levels will be assessed at baseline, on Day 1 of the first two cycles, and a final sample will be collected at progression or end of treatment (whichever comes first). The distribution of levels of serum microRNA will be checked and, if needed, data transformation will be employed for normality. The levels of serum miRNA will be descriptively summarized using differential expression (DE) fold change > 2 p0.05 and 95% CI for each timepoint. The changes in serum miRNA will be also descriptively summarized using the same descriptive statistics. The associations between the change of serum miRNA and each of the efficacy outcomes (OS and PFS) will be descriptively evaluated using logistic and Cox proportional hazard regression models. The proportional hazard assumption will be checked and, if violated, a weighed Cox regression model or restricted mean survival time will be utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Najeeb Al Hallak, MD, Principal Investigator — Wayne State University
Locations (9):
- United States (9):
  - Karmanos Cancer Institute at McLaren Bay Region, Bay City, Michigan
  - Karmanos Cancer Institute at McLaren Clarkston, Clarkston, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute at McLaren Flint, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Karmanos Cancer Institute at McLaren Lapeer Region, Lapeer, Michigan
  - Karmanos Cancer Institute at McLaren Macomb, Macomb, Michigan
  - Karmanos Cancer Institute at McLaren Northern Michigan, Petoskey, Petoskey, Michigan
  - Karmanos Cancer Institute at McLaren Port Huron, Port Huron, Michigan